CLINICAL TRIAL: NCT06399588
Title: Intervention for Adolescent Tobacco Initiation Prevention (IATIP) to Promote Health and Well-being: A Protocol for a Pilot Feasibility Cluster Randomised Controlled Trial in Dhaka, Bangladesh
Brief Title: Intervention for Adolescent Tobacco Initiation Prevention
Acronym: IATIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Commonwealth Scholarship Commission (Unknown)
Responsible Party: Principal Investigator, Sahadat Hossain, Principal Investigator, University College, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22645/004
Record Dates: First submitted 2024-04-26; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Health Behaviour; Tobacco Prevention; Well-being
Keywords: Adolescent; Tobacco initiation; Health and Well-being; Prevention; School-based intervention; C-RCT; Bangladesh
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: This trial will have two groups: intervention and control. The unit of randomisation will be schools, where the adolescents enrolled in school years 8 and 9 in Dhaka, Bangladesh.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention consists of three 40-minute sessions, delivered over three successive days, including knowledge and skill-based lectures, interactive activities, and materials targeting tobacco prevention and health promotion.
  Interventions: Behavioral: Intervention for Adolescent Tobacco Initiation Prevention (IATIP)
- Control group (No Intervention): Participating schools in the control group will maintain their regular ongoing activities without introducing the IATIP. Students in the control group will not receive any specific anti-tobacco or health and well-being promotion materials beyond their standard school curriculum.

INTERVENTIONS:
Behavioral: Intervention for Adolescent Tobacco Initiation Prevention (IATIP) — The IATIP is an evidence-based tobacco prevention program tailored for Bangladeshi adolescents, integrating Behavior Change Techniques, the Behavior Change Wheel, and the Theoretical Domains Framework. Utilizing the Arena Blended Connected (ABC) model ensures effective delivery. Six key learning types are integrated to optimize knowledge acquisition, concept exploration, collaboration, discussions, practical application, and skill development. The curriculum comprises three core components addressing adolescents' challenges: the information curriculum cultivates factual awareness, the social competence curriculum strengthens refusal skills and social competencies, and the social influence curriculum builds resilience against tobacco-promoting social influences.
  Arms: Intervention group

SUMMARY:
This school-based cluster randomized controlled trial aims to assess the feasibility of implementing the Adolescent Tobacco Initiation Prevention (IATIP) and evaluate the potential efficacy of IATIP in preventing tobacco initiation and promoting the health and well-being of school adolescents in Dhaka, Bangladesh. The intervention consists of three 40-minute sessions, delivered over three successive days, including knowledge and skill-based lectures, interactive activities, and materials targeting tobacco prevention and health promotion.

DETAILED DESCRIPTION:
Background and Aims: Adolescent tobacco use is a significant public health challenge, particularly in low- and middle-income countries like Bangladesh. An Intervention for Adolescent Tobacco Initiation Prevention (IATIP) has been developed to address this issue. This study aims to assess the feasibility of implementing the IATIP and evaluate its potential efficacy in preventing tobacco initiation and promoting health and well-being.

Design: Pilot feasibility school-based cluster randomized controlled trial.

Setting: Secondary schools in Dhaka city, Bangladesh.

Participants: Adolescents in school years 8 and 9 attending participating schools in Dhaka (K = 8 clusters; N~1280 participants).

Intervention: The intervention consists of three 40-minute sessions, delivered over three successive days, including knowledge and skill-based lectures, interactive activities, and materials targeting tobacco prevention and health promotion. This intervention was developed based on evidence gathered from a quantitative survey, qualitative focus groups, and a systematic review.

Measurements: The primary outcome is the feasibility of the intervention, assessed with recruitment and attrition rates, fidelity of delivery and acceptability. Secondary outcomes include the change in intention to initiate tobacco use; tobacco knowledge, attitudes, and beliefs; skills development related to tobacco resistance; and the promotion of mental well-being. Data will be collected through structured questionnaires administered at baseline and 1-month follow-up assessments for both intervention and control groups. A post-intervention process evaluation will be conducted among the students who participated in the intervention and the teachers using a mixed-method approach, incorporating both questionnaires and semi-structured interviews, to gain insights into intervention implementation, facilitation, participant experiences, and identify potential areas for improvement.

Comments: This pilot feasibility trial addresses a critical gap in tobacco prevention initiatives tailored for Bangladeshi school adolescents. By combining evidence-based strategies, IATIP aims to empower adolescents with the knowledge and skills needed to resist tobacco initiation, while also targeting specific components to improve health and well-being, recognising the interconnected challenges of tobacco use and health and well-being among adolescents. Successful implementation of this pilot trial has the potential to reduce the intention to initiate tobacco use, limit exposure to second-hand smoke, and contribute to the overall health and well-being of school adolescents. Given the scalability of school-based interventions, the trial's success may pave the way for future large-scale definitive trials, influencing national policies and strategies.

ELIGIBILITY:
Inclusion Criteria:

* Bangladeshi school adolescent
* Students at one of the participating schools
* Students of Years 8 and 9

Exclusion Criteria:

* Students of physical and mental impairment
* don't understand and read the 'Bangla' language
* don't have parental consent

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1280 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention: recruitment rate | Before starting the intervention, an average of 10 days.
  The percentage of eligible participants who agree to take part in the study will be calculated to evaluate recruitment rate.
Feasibility of the intervention: attrition rate | Through study completion, an average of 2 months.
  The dropout rate will be monitored as a measure of attrition, specifically, calculating the percentage of recruited participants who do not complete the follow-up assessment.
Feasibility of the intervention: fidelity of delivery | Immediately after the completion of the intervention delivery, an average of 30 days.
  The fidelity of intervention delivery will be assessed using a pre-defined index, consisting of 21 content items. A 3-point Likert (0 = not implemented, 1 = partially implemented and 2 = fully implemented) will be used to assess the fidelity index. A higher score indicates a more fidelity of intervention delivery.
Feasibility of the intervention: acceptability | Immediately after the completion of the intervention delivery, an average of 30 days.
  To evaluate the acceptability of the intervention, participants' perceptions of the intervention's relevance, and appropriateness will be explored. Participants will be asked a 5-point Likert scale question: "To what extent do you feel the study sessions met your expectations?", with response options ranging from 1 (not at all) to 5 (completely). They will also be asked, "To what extent do you think the components were relevant to preventing tobacco initiation and promoting health and well-being?" and "To what extent do you think the images and videos presented in the sessions were appropriate and relevant to the contents?" with the same measures. The clarity and comprehensibility of the intervention materials, such as handbooks and presentations, will be rated on a 5-point Likert scale from 1 (not at all) to 5 (extremely). A higher score indicates a more acceptable intervention.

SECONDARY OUTCOMES:
Change in the intention to initiate tobacco use | Up to 5 weeks
  To assess this, a two-item Likert scale will be used: (1) "if someone (cousin/friend/close relative) offers you a tobacco product, would you use it?" and (2) "at any time during the next 12 months, do you think you will use any form of tobacco?". Responses to these questions will be categorized into four options: "Definitely not," "Probably not," "Probably yes," and "Definitely yes." This scale produces a potential range of 0-6, with lower scores indicating a lower likelihood of intending to initiate tobacco use within the next 12 months. The potential effect of the intervention will be determined by changes in scores between baseline and follow-up.
Change in self-rated physical health score | Up to 5 weeks
  To assess self-rated physical health status, participants will be asked to rate their overall physical health conditions with five response options: 1 = very poor, 2 = poor, 3 =moderate, 4 = good and 5 = very good. The response options will be treated as a continuous ordinal measure. Therefore, a higher score indicates a better health condition. The potential effect of the intervention will be determined by changes in scores between baseline and follow-up.
Evaluate the promotion of overall mental well-being | Up to 5 weeks
  The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) will be used to measure participants' overall mental well-being. This validated 7-item 5-point Likert scale scores range from 7 to 35 and higher scores indicate higher positive mental wellbeing. The potential effect of the intervention will be determined by changes in scores between baseline and follow-up.
Change in stress score | Up to 5 weeks
  To assess the participants' level of stress, the 10-item Perceived Stress Scale (PSS) will be used. This widely recognized scale assesses the extent to which individuals perceive situations in their lives as stressful. Responses will be collected on a 5-point Likert scale, with 0 indicating 'never,' 1 = almost never, 2 = sometimes, 3 = fairly often, and 4 indicating 'very often.' A total score for each adolescent will be obtained by summing the scores across all 10 items for a total range of 0 to 40. A higher score indicates higher perceived stress. The potential effect of the intervention will be determined by changes in scores between baseline and follow-up.
Change in anxiety score | Up to 5 weeks
  One of the most popularly used 7-item scales, the Generalized Anxiety Disorder-7 (GAD-7) will be used to identify participant's anxiety in this trial. Participants will be asked how often they were bothered by each of the seven core symptoms of GAD with four response options: 0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day, over the last 14 days. The response options will also be calculated as a continuous ordinal measure. Therefore, the range of scores of the GAD-7 will be 0 to 21. A higher score indicates a higher level of anxiety. The potential effect of the intervention will be determined by changes in scores between baseline and follow-up.
Change in depression score | Up to 5 weeks
  The Patient Health Questionnaire-9 (PHQ-9) will be used to assess the level of depression. Participants will be asked how often they were bothered by each of the nine core symptoms of PHQ-9 with four response options: 0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day, over the last 14 days. The response options will also be calculated as a continuous ordinal measure. Therefore, the range of scores of the GAD-7 will be 0 to 27. A higher score indicates a higher level of depression. The potential effect of the intervention will be determined by changes in scores between baseline and follow-up.
Change in knowledge | Up to 5 weeks
  To assess participant's knowledge about tobacco and health, a set of 20 items will be used. A participant will earn 1 point for each correct response, while an incorrect or unknown answer will be scored as 0 points. The cumulative knowledge score will be calculated by summing the points from all items, with a maximum achievable score of 20 points. A higher score indicates a more knowledgeable individual. The potential effect of the intervention will be determined by changes in scores between baseline and follow-up.
Change in attitudes | Up to 5 weeks
  To measure participants' attitudes toward tobacco and health, a 16-item standardized scale will be utilised. Each item is structured as a Likert-type scale with five ranks. A quantitative approach will be employed to summarize the responses across all attitude items. For positive attitude items, responses of ''extremely agree'' will be scored as 5 points, ''agree'' as 4 points, ''unclear'' as 3 points, ''disagree'' as 2 points, and ''extremely disagree'' as 1 point. Conversely, for negative attitude items, the scoring will be reversed as 1, 2, 3, 4, and 5 points. The total attitude scale score will be the sum of all item scores, with a maximum attainable score of 80 points and a minimum of 16 points. A higher score indicates a more negative attitude toward tobacco.
Change in beliefs | Up to 5 weeks
  To assess participants' beliefs about tobacco use, an 8-item scale will be used. This scale focuses on both positive (4 items) and negative (4 items) beliefs concerning various aspects of tobacco use. Participants will be asked to rate the likelihood of each scenario happening to them if they use tobacco in the next month. Responses will be collected on a 4-point Likert-type scale: 1=very likely, 2=likely, 3=unlikely, 4=very unlikely. Positive beliefs (score 8 to 32) include feeling relaxed, having fun, being popular, and being confident and outgoing. Negative beliefs (score 8 to 32) encompass issues with parents and friends, financial problems, and the risk of addiction. A lower score indicates more positive or negative beliefs about tobacco.
Skill development: Decision-making | Up to 5 weeks
  For 'Decision-Making Skills,' Participants will respond to statements reflecting different approaches to decision-making, indicating their level of agreement (1=Strongly Agree, 2=Agree, 3=Disagree, 4=Strongly Disagree) across five items. Differences in item responses between baseline and follow-up will be assessed to evaluate the effect of the intervention.
Skill development: Refusal skill | Up to 5 weeks
  For 'Refusal Skills,' participants will navigate hypothetical situations, expressing their likelihood of refusal (1=Very Likely, 2=Likely, 3=Unlikely, 4=Very Unlikely) in response to three scenarios. Differences in item responses between baseline and follow-up will be assessed to evaluate the effect of the intervention.
Skill development: Self-esteem | Up to 5 weeks
  'Self-esteem' will be assessed through agreement with self-descriptive statements (1=Strongly Agree, 2=Agree, 3=Disagree, 4=Strongly Disagree), encompassing ten items. Differences in item responses between baseline and follow-up will be assessed to evaluate the effect of the intervention.
Skill development: Problem solving | Up to 5 weeks
  'Problem-Solving Skills' will be assessed by responses to statements related to interpersonal dealings (1=Strongly Agree, 2=Agree, 3=Disagree, 4=Strongly Disagree), consisting of five items. Differences in item responses between baseline and follow-up will be assessed to evaluate the effect of the intervention.
Skill development: Assertiveness | Up to 5 weeks
  'Assertiveness' will be evaluated by considering the ease or difficulty participants perceived in accomplishing certain tasks (1=Very Easy, 2=Easy, 3=Difficult, 4=Very Difficult) across six scenarios. Differences in item responses between baseline and follow-up will be assessed to evaluate the effect of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sahadat Hossain, MSPH, Principal Investigator — University College, London
Locations (1):
- Secondary schools, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
We will not release any identifiable data of the participants to any third parties, in accordance with our ethical obligations. However, the overall anonymized dataset will be made available upon request, solely for research purposes.

REFERENCES:
- [Derived] Hossain S, Beard E, Shahab L. Intervention for adolescent tobacco initiation prevention (IATIP) to promote health and well-being: a protocol for a pilot cluster randomised controlled trial in Dhaka, Bangladesh. Pilot Feasibility Stud. 2025 Nov 17;11(1):145. doi: 10.1186/s40814-025-01710-9. PMID 41250156